CLINICAL TRIAL: NCT06006689
Title: A Randomized, Double-blind, Multi-center, Standardise-loaded, Placebo-parallel Controlled Clinical Trial of Efficacy and Safety of QiShen YiQi Dripping Pills in the Treatment of Diabetic Kidney Disease (Syndrome of Qi Deficiency With Blood Stasis)
Brief Title: Efficacy and Safety of QiShen YiQi Dripping Pills in the Treatment of Diabetic Kidney Disease (Syndrome of Qi Deficiency With Blood Stasis)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-QSYQDW-DKD-Ⅱ
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Qishen Yiqi Dripping Pills placebo, 3 bags, take orally after meals, 3 times a day
  Interventions: Drug: Qishen Yiqi Dripping Pills placebo 3 bags
- Low dose group (Experimental): Low dose Qishen Yiqi Dripping Pills, 3 bags, take orally after meals, 3 times a day
  Interventions: Drug: Low dose Qishen Yiqi Dripping Pills 3 bags
- High dose group (Experimental): High dose Qishen Yiqi Dripping Pills, 3 bags, take orally after meals, 3 times a day
  Interventions: Drug: High dose Qishen Yiqi Dripping Pills 3 bags

INTERVENTIONS:
Drug: Qishen Yiqi Dripping Pills placebo 3 bags — Qishen Yiqi Dripping Pills placebo contain Qishen Yiqi dripping pills placebo 3 bags(0.52g dripping pills placebo per bag),take orally after meals, 3 times a day for 12weeks
  Other Names: Placebo group
  Arms: Placebo group
Drug: Low dose Qishen Yiqi Dripping Pills 3 bags — Low dose Qishen Yiqi Dripping Pills contain Qishen Yiqi dripping pills 2 bags(0.52g dripping pills per bag) and Qishen Yiqi dripping pills placebo 1 bag(0.52g dripping pills placebo per bag),take orally after meals, 3 times a day for 12weeks
  Other Names: Low dose group
  Arms: Low dose group
Drug: High dose Qishen Yiqi Dripping Pills 3 bags — High dose Qishen Yiqi Dripping Pills contain Qishen Yiqi dripping pills 3 bags(0.52g dripping pills per bag),take orally after meals, 3 times a day for 12weeks
  Other Names: High dose group
  Arms: High dose group

SUMMARY:
This study will evaluate the efficacy and Safety of QiShen YiQi Dripping Pills in the treatment of Diabetic Kidney Disease (syndrome of Qi deficiency with blood stasis)

ELIGIBILITY:
Inclusion Criteria:

* Man or woman between 18-75 years-old
* Subjects with type 2 diabetes mellitus
* Subjects with a clinical diagnosis of diabetic kidney disease
* eGFR≥ 45 mL/min/1.73 m2
* UACR ≥ 30 mg/g but ≤ 300 mg/g
* Conformed to the TCM syndrome differentiation standard of chronic heart failure syndrome of Qi deficiency and blood stasis
* Received Steady dose of ACEI or ARB therapy for chronic heart failure at least 2 weeks before receiving investigational drug
* Abide by the experimental protocol and cooperate with the data collection according to the researcher's judgment

Exclusion Criteria:

* Subjects with type 1 diabetes mellitus or other specific types of diabetes
* Acute complications of diabetes such as diabetic ketoacidosis and hyperosmolar hyperglycemia occurred in the past 3 months
* HbA1c ≥8.5% or fasting blood glucose >11 mmol/L
* Urinary sediment indicates "active" glomerulogenic hematuria
* Subjects have been clinically confirmed cases of primary glomerular disease, secondary glomerular disease other than DKD or other systemic diseases
* The presence of uncontrolled hypertension, systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg or Hypotension with a systolic blood pressure <90mmHg and/or a diastolic blood pressure <60mmHg
* ALT or AST> 2 times the upper limit of normal
* Serum potassium> the upper limit of normal
* Patients with unstable basic treatment for lowering blood glucose and blood lipids within the past 3 months, and patients with unstable basic treatment for lowering blood pressure within the past 1 month (changing the type of drugs, such as changing the β-receptor blockers to calcium ion antagonists, etc.)
* Take the following medications within the last 2 weeks：a. Other drugs for the treatment of DKD (Finerenone, Keluoxin capsule, Qizhi Yishen capsule, SGLT2i drugs, GLP-1 drugs, etc.), b. Calcium oxybenzenesulfonate for the treatment of diabetic retinopathy, c. Chinese patent medicine, Chinese medicine decoction, formula granule and other Chinese medicine preparations with the same composition or function indications, d. Tripterygium wilfordii related preparations, Huangkui capsule
* Patients who need to take antiplatelet drugs, the dose was stable for less than 1 month
* Serious diseases of other systemic systems that may affect the judgment of efficacy and safety
* A history of alcohol or drug abuse with a combination of mental illness and poor control
* Allergic to the experimental drug or its ingredients
* Women who are pregnant or breastfeeding, or who have a need to have children during the trial
* Participating in other clinical studies and taking investigational drugs from other studies within 3 months prior to screening
* The investigator deems that the patient is not suitable to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in UACR(urinary albumin ⁃ to ⁃ creatinine ratio). | Baseline to weeks 4, 8 and 12
  Change in UACR from baseline to weeks 4, 8 and 12.

SECONDARY OUTCOMES:
Ratio of subjects with UACR returned to normal. | Baseline to weeks 4, 8 and 12
  Ratio of subjects with UACR returned to normal at weeks 4, 8 and 12.
Ratio of subjects with UACR decrease of more than 30% from baseline. | Baseline to weeks 4, 8 and 12
  Ratio of subjects with UACR decrease of more than 30% from baseline at weeks 4, 8 and 12.
Ratio of subjects from microalbuminuria stage to macroalbuminuria | Baseline to weeks 4, 8 and 12
  Ratio of subjects from microalbuminuria stage to macroalbuminuria at weeks 4, 8 and 12.
Change in eGFR(estimated glomerular filtration rate). | Baseline to weeks 4, 8 and 12
  Change in eGFR from baseline to weeks 4, 8 and 12.
Change in Traditional Chinese Medicine Syndrome Score | Baseline to weeks 4, 8 and 12
  Change in Traditional Chinese Medicine Syndrome Score from baseline to weeks 4, 8 and 12. There were 9 clinical primary symptoms, 7 clinical secondary symptoms, tongue picture and pulse condition evaluated as TCM symptoms, which was defined as TCM syndrome score. The standard of TCM primary symptoms and secondary symptoms scored as without 0, light 2, medium 4, heavy 6 points. Tongue picture and pulse condition did not count.
TCM syndrome | Baseline to weeks 4, 8 and 12
  Number and ratio of subjects with Clinical recovery, obvious effect, effective or ineffective in curative effect of TCM syndrome at weeks 4, 8 and 12.

OTHER OUTCOMES:
Change in β2-MG. | Baseline to weeks 4, 8 and 12
  Change in β2-MG from baseline to weeks 4, 8 and 12.
Change in Cys-C. | Baseline to weeks 4, 8 and 12
  Change in Cys-C from baseline to weeks 4, 8 and 12.
Change in PCX. | Baseline to week 12
  Change in PCX from baseline to week 12.
Change in MCP-1. | Baseline to week 12
  Change in MCP-1 from baseline to week 12.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - Dongzhimen Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - The Affiliated TCM Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Hebei Province Hospital of Traditional Chinese Medicine, Shijiazhuang, Hebei
  - Heilongjiang Academy of Traditional Chinese Medicine (Heilongjiang Provincial Hospital of Traditional Chinese Medicine), Harbin, Heilongjiang
  - Kaifeng Hospital of Traditional Chinese Medicine, Kaifeng, Henan
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - Shananxi Province Hospital of Traditional Chinese Medicine, Xi'an, Shananxi
  - Longhua Hospital affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality
  - Hangzhou hospital of traditional Chinese medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang